CLINICAL TRIAL: NCT06000111
Title: Duration of Face Down Positioning Following Full-Thickness Macular Hole Repair: a Randomized Feasibility Study
Brief Title: Duration of Face Down Positioning for Full-Thickness Macular Hole Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Varun Chaudhary, Professor, Department of Surgery, Chief of Ophthalmology, Hamilton Regional Eye Institute, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16100
Record Dates: First submitted 2023-07-24; First posted 2023-08-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Intervention Model Description: This study will be a single-centered, parallel group randomized controlled feasibility trial. Patients will be randomized 1:1 between groups.
Who Masked: Outcomes Assessor
Masking Description: The surgeon will be masked to the patient's treatment allocation until after surgery is complete. At this point, the surgeon will be made aware of the patient's treatment allocation and inform the patient in the recovery room regarding their treatment allocation. The participants and the clinical teams managing the patient care will be unmasked. The outcome assessors will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Face-Down Positioning for 3-Days and Nights (Experimental): Patients allocated to this study arm will maintain face-down positioning for 3-days and nights post-operatively. Patients will be advised to posture immediately following surgery and will be advised to posture for 50 minutes of each hour. Patients will be advised that during their 10-minute break each hour, they should avoid face-up positioning. FDP will be advised during both waking and sleeping hours.
  Interventions: Behavioral: 3 Days of face-down positioning
- Face-Down Positioning for 7-Days and Nights (Active Comparator): Patients allocated to this study arm will maintain face-down positioning for 7-days and nights post-operatively. Patients will be advised to posture immediately following surgery and will be advised to posture for 50 minutes of each hour. Patients will be advised that during their 10-minute break each hour, they should avoid face-up positioning. FDP will be advised during both waking and sleeping hours.
  Interventions: Behavioral: 7 Days of face-down positioning

INTERVENTIONS:
Behavioral: 3 Days of face-down positioning — Following surgical repair, patients in the intervention group will maintain 3-days and nights of face-down positioning post-operatively.
  Arms: Face-Down Positioning for 3-Days and Nights
Behavioral: 7 Days of face-down positioning — Following surgical repair, patients in the intervention group will maintain 7-days and nights of face-down positioning post-operatively.
  Arms: Face-Down Positioning for 7-Days and Nights

SUMMARY:
A full-thickness macular hole is when there is a small gap that opens in the center part of the retina (the light-sensitive layer of tissue in the back of the eye). Following surgical repair of these holes, patients have to lie face down for a number of days and nights. The exact amount of time necessary to position is however unknown. The goal of this randomized feasibility clinical trial is to compare 3 days and nights of face-down positioning to 7 days and nights of face-down positioning following pars plana vitrectomy surgery for full-thickness macular holes on key patient outcomes. This study will be a feasibility study to better inform a future larger clinical trial. Additionally, this investigation will be examining the rates of macular hole closure, patient visual acuity following surgery, patient quality of life, patient compliance, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with an idiopathic full-thickness macular hole
* Symptom duration of less than 6 months
* Patient must agree to participate in this investigation

Exclusion Criteria:

* Macular hole minimum diameter >1000 μm
* A history of high myopia (> -6)
* Traumatic macular hole
* Amblyopia
* Retinal vein occlusion
* Inflammatory eye diseases
* Patients found to have a retinal tear during either the pre-operative assessment or intraoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | The recruitment rate will be calculated during the recruitment period.
  This investigation's primary objective will be focused on assessing feasibility. One primary outcome will be to evaluate the recruitment rate of this study.
Retention Rate | The retention rate will be calculated at 3-months post-operatively.
  This investigation's primary objective will be focused on assessing feasibility. One primary outcome will be to evaluate the retention rate of this study.
Completion Rate | The completion rate will be calculated at 3-months post-operatively.
  This investigation's primary objective will be focused on assessing feasibility. One primary outcome will be to evaluate the completion rate of this study.
Recruitment Time | The recruitment time will be calculated during the recruitment period.
  This investigation's primary objective will be focused on assessing feasibility. One primary outcome will be to evaluate the recruitment time for this study.

SECONDARY OUTCOMES:
Macular Hole Closure Rate | 3-months post-operatively
  The rate of macular hole closure will be evaluated by 2-independent readers masked to treatment allocation. They will grade the outcome as open or closed. Outcomes classified as open will be further divided into open and flat (without a cuff of subretinal fluid) or open and elevated (with a cuff of subretinal fluid).
Best-Corrected Visual Acuity (BCVA) | 3-months post-operatively
  Patient best-corrected visual acuity will be measured by Snellen visual acuity. With this measure of visual acuity, visual acuity can range from 20/10 (best) to 20/1000 (worst). If the patient is unable to read the chart at any distance, patients will next be assessed whether they can count figures at a given distance, if not, they will be tested to see whether they can perceive hand motion and if not, if they can perceive any light.
Vision specific quality of life measure | 3-months post-operatively
  The National Eye Institute Visual Function Questionnaire (NEI VFQ-25) will be administered to patients. Possible patient scores range from 0 to 100 with a higher score representing higher vision-related quality of life.
Compliance with Face Down Positioning | While the patient is positioning; this will either be for 3 days or 7 days depending on their treatment allocation.
  Compliance will be assessed with self-administered questionnaires assessing the patients' compliance during the morning, midday, evening, and overnight. The possible range of scores is from 1 to 10 with higher scores indicating better compliance.
Complication Rates | Rates will be determined for the entire follow-up period (3-months)
  Specifically, the rates of endophthalmitis, retinal detachment, and vitreous hemorrhage
Health Related Quality of Life Measure | 3-months post-operatively
  The Quality of Life Scale (QOLS) will be administered to patients. The range of possible patient scores is from 16 to 112. Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Varun Chaudhary, MD, FRCSC, Principal Investigator — McMaster University, St. Joseph's Hospital
Locations (1):
- St. Joseph's Hospital King Campus, Stoney Creek, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be shared with other researchers upon reasonable request.

REFERENCES:
- [Derived] Nanji K, Oquendo PL, Srinivasan S, Vyas C, Prasad F, Farrokhyar F, Chaudhary V. Duration of face down positioning following full-thickness macular hole repair: A protocol for a randomized pilot study. PLoS One. 2024 Aug 20;19(8):e0304566. doi: 10.1371/journal.pone.0304566. eCollection 2024. PMID 39163327